CLINICAL TRIAL: NCT04094285
Title: The Effect of Hyperoxia and Hypoxia on Fluorescence Lifetime Imaging Ophthalmoscopy in Healthy Subjects- a Randomized, Double Blind, Crossover Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD. Dr. med. univ., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-070119
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: To Investigate the Effect of 100% Oxygen Breathing on Fluorescence Lifetime Imaging Ophthalmoscopy (FLIO) in Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: SAUERSTOFF; Drug: STICKSTOFF
- 2 (Experimental)
  Interventions: Drug: SAUERSTOFF; Drug: STICKSTOFF

INTERVENTIONS:
Drug: SAUERSTOFF — SAUERSTOFF medizinisch, Messer GmbH, Industriestrasse 5, 2352 Gumpoldskirchen, Austria
  Dose:
  min. 95.5%, breathing for 30 minutes
Drug: STICKSTOFF — STICKSTOFF medizinisch, Messer GmbH, Industriestrasse 5, 2352 Gumpoldskirchen, Austria
  Dose:
  88% with 12% oxygen, breathing for 30 minutes

SUMMARY:
The present study aims to investigate whether FLIO can also detect shorttime changes in retinal metabolism induced by hyperoxia and hypoxia. For this purpose, 48 healthy subjects will be included in the present study and changes in FLIO will be assessed during breathing of 100% oxygen to induce hyperoxia as well as during breathing of 12% oxygen in nitrogen to induce hypoxia. Since stimulation with flickering light also induces a higher metabolic demand in the retina (functional hyperemia), thisprovocation test will also applied during breathing of the different gas mixtures and compared to baseline. To gain information about retinal blood flow, optical coherence tomography angiography (OCT-A) will be performed. The results of the present study can help to gain more insight into the physiology of the retinal metabolism and might give grounds to establish new biomarkers in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years

  * Normal ophthalmic findings
  * Ametropia ≤ 6 diopters
  * Normal findings in the medical history and physical examination including ECG unless the investigator considers an abnormality to be clinically irrelevant
  * Nonsmokers

Exclusion Criteria:

Regular use of medication, abuse of alcoholic beverages or drugs

* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* History or family history of epilepsy
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in FLIO induced by hyperoxia | 15 minutes

SECONDARY OUTCOMES:
Changes in FLIO induced by hypoxia | 15 minutes
Changes in FLIO induced by flicker stimulation | 15 minutes
Changes in OCT-A induced by hyperoxia | 15 minutes
Changes in OCT-A induced by hypoxia | 15 minutes
Changes in OCT-A induced by flicker stimulation | 15 minutes
Retinal oxygen saturation | 15 minutes
Retinal vessel diameter | 15 minutes
Changes in peripheral oxygen saturation | 15 minutes
Changes in blood gas parameters (pH, pCO2, PO2 and SaO2) | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Austria, Vienna, Austria

REFERENCES:
- [Derived] Pai V, Janku P, Lindner T, Graf U, Schmetterer L, Garhofer G, Schmidl D. A New Approach to Retinal Oxygen Extraction Measurement Based on Laser Speckle Flowgraphy and Retinal Oximetry. Transl Vis Sci Technol. 2024 Dec 2;13(12):12. doi: 10.1167/tvst.13.12.12. PMID 39661379